CLINICAL TRIAL: NCT00530712
Title: The US StuDy for EvalUating EndovasculaR TreAtments of Lesions in the Superficial Femoral Artery and Proximal Popliteal By usIng the Protege EverfLex NitInol STent SYstem II
Brief Title: Safety and Effectiveness Study of EverFlex Stent to Treat Symptomatic Femoral-popliteal Atherosclerosis
Acronym: DURABILITY II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-2424
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Peripheral Vascular Diseases; Claudication
Keywords: SFA; Popliteal; Stent; EverFlex
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PTA and Stenting with EverFlex device (Experimental): Qualified subjects undergo treatment of atherosclerotic lesions in the native SFA/SFA/PPA with PTA and stenting using the PROTÉGÉ® EverFlex™ Self-Expanding Stent System
  Interventions: Device: PROTÉGÉ® EverFlex™ Self-Expanding Stent System

INTERVENTIONS:
Device: PROTÉGÉ® EverFlex™ Self-Expanding Stent System — Implantation of a single study device in the native superficial femoral artery or superficial femoral artery and proximal popliteal artery.

SUMMARY:
This is a multi-center, non-randomized, single arm study to compare PTA and primary stenting using a single PROTÉGÉ® EverFlex™ stent to performance goals of PTA alone in the treatment of atherosclerotic superficial femoral artery (SFA) and proximal popliteal lesions.

ELIGIBILITY:
Inclusion Criteria:

* Stenotic, restenotic (from PTA or adjunct therapy, not including stents or stent grafts) or occluded lesion(s) located in the native superficial femoral artery or superficial femoral and proximal popliteal arteries.
* Symptomatic femoral-popliteal atherosclerosis.
* Willing to comply with all follow-up evaluations at the specified times.
* Provides written informed consent prior to enrollment in the study.

Exclusion Criteria:

* Previously implanted stent(s) or stent graft(s) in the target vessel.
* Planned use of devices other than angioplasty balloons during procedure.
* Received endovascular treatment of the target lesion (except stents/stent grafts) within six months of the index procedure.
* Life expectancy of less than 12 months.
* Symptomatic femoral disease in the opposite limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2007-08; Primary Completion 2012-03 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Matsumura, MD, Principal Investigator — University of Wisconsin, Madison; Krishna Rocha-Singh, MD, Principal Investigator — Prairie Heart Institute

REFERENCES:
- [Result] Matsumura JS, Yamanouchi D, Goldstein JA, Pollock CW, Bosiers M, Schultz GA, Scheinert D, Rocha-Singh KJ. The United States StuDy for EvalUating EndovasculaR TreAtments of Lesions in the Superficial Femoral Artery and Proximal Popliteal By usIng the Protege EverfLex NitInol STent SYstem II (DURABILITY II). J Vasc Surg. 2013 Jul;58(1):73-83.e1. doi: 10.1016/j.jvs.2012.12.066. Epub 2013 May 2. PMID 23642924

RESULTS

PARTICIPANT FLOW:
Groups:
- EverFlex™ Peripheral Self-Expanding Stent System: Subjects recieved the EverFlex™ Peripheral Self-Expanding Stent System
Period: Enrollment
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Started | 287 (Total Enrolled Subjects)
Completed | 287 (Subjects Available at Discharge)
Not Completed | 0
Period: 30 Day Follow-up Visit
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Started | 287 (Subjects Expected for 30-Day Visit)
Completed | 280 (Subjects that Completed 30-Day Follow-up Visit)
Not Completed | 7
Not completed — Withdrawal by Subject | 2
Not completed — Missed Visit | 5
Period: 6 Month Follow-up Visit
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Started | 287 (Subjects Expected for 6-Month Visit)
Completed | 275 (Subjects that Completed 6-Month Follow-up Visit)
Not Completed | 12
Not completed — Withdrawal by Subject | 4
Not completed — Missed Visit | 3
Not completed — Lost to Follow-up | 3
Not completed — Death | 2
Period: 12 Month Follow-up Visit
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Started | 287 (Subjects Expected for 12 Month Visit)
Completed | 263 (Subjects that Completed 12-Month Follow-up Visit)
Not Completed | 24
Not completed — Withdrawal by Subject | 5
Not completed — Missed Visit | 3
Not completed — Lost to Follow-up | 7
Not completed — Death | 9

BASELINE CHARACTERISTICS:
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 190
Region of Enrollment [Number; unit: participants]
  United States | 244
  Europe | 43

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency
Description: Primary stent patency, as determined by the core laboratory, was defined as PSV ratio < 2.0 at the stented target lesion as measured by duplex ultrasound at the 1-year follow-up visit (335-395 days post procedure) and no clinically-driven TLR within the stented segment within 1 year of the procedure.
Time Frame: 1 Year
Measure: Number; unit: Percentage of participants with data
Groups:
- EverFlex™ Peripheral Self-Expanding Stent System: Subjects recieved the EverFlex Peripheral Self-Expanding Stent
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 226
Percentage of participants with data | 67.7

2. Primary Outcome: Major Adverse Events
Description: Major Adverse Events (MAE) was defined as clinically-driven Target Lesion Revascularization (TLR), amputation of treated limb, or all-cause mortality, as adjudicated by the Clinical Events Commettee (CEC)
Time Frame: 30 Days
Measure: Number; unit: Percentage of participants with data
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 284
Percentage of participants with data | 0

3. Secondary Outcome: Single-Stent Primary Patency
Description: Primary stent patency in subjects with single-stent, as determined by the core laboratory, was defined as PSV ratio < 2.0 at the stented target lesion as measured by duplex ultrasound at the 1-year follow-up visit (335-395 days post procedure) and no clinically-driven TLR within the stented segment within 1 year of the procedure. Single stents were implanted in 272 subject.
Time Frame: 1 Year
Measure: Number; unit: Percentage of participants with data
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 217
Percentage of participants with data | 68.7

4. Secondary Outcome: Single-Stent Major Adverse Events
Description: MAE rate in subjects who received a single stent was defined as clinically-driven TLR, amputation of treated limb, or all-cause mortality that occurred within 30-days post-procedure, as adjudicated by the CEC. Single stents were implanted in 272 subjects.
Time Frame: 30 Days
Measure: Number; unit: Percentage of participants with data
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 270
Percentage of participants with data | 0

5. Secondary Outcome: Major Adverse Events
Description: MAE rate at 1 year was defined as clinically-driven TLR, amputation of treated limb, or all-cause mortality that occurs within 1 year post-procedure, as adjudicated by the CEC.
Time Frame: 1 Year
Measure: Number; unit: Percentage of particants with data
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 273
Percentage of particants with data
  Subjects with MAE | 16.8
  Death | 2.9
  Amputation | 0
  Clinically-driven TLR | 13.9

6. Secondary Outcome: Stent Fracture Rate
Description: Stent integrity determined by x-ray at 1, 2 and 3 years post stent implantation.
Time Frame: 1, 2 and 3 Years
Population: 263 stents analyzable at 1 year
Measure: Number; unit: percentage of stents implanted
Units Other Than Participants: Stent Implanted
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 251
Number analyzed (Stent Implanted) | 263
percentage of stents implanted
  1 year | 0.4
  2 year: number analyzed (Participants) | 214
  2 year: number analyzed (Stent Implanted) | 226
  2 year | 1
  3 year: number analyzed (Participants) | 207
  3 year: number analyzed (Stent Implanted) | 217
  3 year | 0

7. Secondary Outcome: Number of Participants With Decline in Rutherford Clinical Category
Description: Defined as an increase of one or more categories in Rutherford Clinical classification compared to baseline. The symptomatic classification is a scale of 0-6, asymptomatic to major tissue loss.
Time Frame: 30 days
Population: Subjects with available RCC data
Measure: Count of Participants; unit: Participants
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 262
Participants | 0

8. Secondary Outcome: Improvement in Rutherford Clinical Category
Description: Improvement in Rutherford Clinical Category (RCC) was defined as an improvement in clinical status indicated by a decrease of one or more categories in RCC compared to baseline.
Time Frame: 1 year
Measure: Number; unit: Percentage of participants with data
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 261
Percentage of participants with data | 83.6

9. Secondary Outcome: Increase in Ankle-Brachial Index From Baseline to 1 Year
Description: Defined as an increase in ancle-brachial index (ABI) at 1 year compared to baseline in subjects with compressible arteries and baseline ABI < 0.9.
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 246
Ratio
  Baseline | 0.65 (0.15)
  1 Year | 0.89 (0.20)

10. Secondary Outcome: Assisted Primary Patency
Description: Assisted primary patency at 1 year was defined as PSV ratio < 2.0 as measured by binary duplex ultrasound maintained by repeated percutaneous intervention completed prior to complete vessel closure. Kaplan-Meier assisted primary patency was evaluated in all enrolled subjects.
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Event free percentage
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 287
Event free percentage | 86.9 [82.1 to 90.4]

11. Secondary Outcome: Secondary Patency
Description: Secondary patency was defined as PSV ratio < 2.0 maintained by repeat percutaneous intervention after occlusion of the target lesion. Secondary patency was evaluated by the Kaplan-Meier method in all enrolled subjects.
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Event free percentage
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 287
Event free percentage | 87.3 [82.6 to 90.8]

12. Secondary Outcome: Absolute Claudication Distance Improvement
Description: Absolute claudication distance improvement at 1 year was defined as the increase in walking distance determined by a graded treadmill exercise test. Only assessed in subjects enrolled under study procol versions in which the endpoint was predefined.
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: Miles
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 74
Miles
  Baseline | 0.23 (0.18)
  1 Year | 0.28 (0.34)

13. Secondary Outcome: Walking Improvement
Description: Walking improvement was defined as an increase in Walking Impairment Questionnaire (WIQ) score in subjects who did not have iliac disease treated at the time of the index procedure compared to baseline.
Time Frame: 1 Year
Population: Subjects with available WIQ data at 1 year
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 241
percent change | 36.8 (40.3)

14. Secondary Outcome: Duplex Ultrasound ≤ 2.4 Primary Patency
Description: Defined as a binary duplex ultrasound ratio ≤ 2.4 at the stented target lesion with no clinically-driven reintervention without the stented segment. Duplex Ultrasound ≤ 2.4 primary patency was evaluated by the Kaplan-Meier method in all enrolled subjects.
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Event free percentage
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 287
Event free percentage | 77.9 [72.4 to 82.4]

ADVERSE EVENTS:
Arm/Group | EverFlex™ Peripheral Self-Expanding Stent System
Serious Adverse Events (participants affected / at risk) | 99/287
Other Adverse Events (participants affected / at risk) | 229/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EverFlex™ Peripheral Self-Expanding Stent System (N=287)
Access site complication - Hematoma (General disorders) | 1
Access site complication - Pseudoaneurysm (General disorders) | 4
Acute Stent Thrombosis (General disorders) | 6
Allergic reaction to contrast dye (General disorders) | 1
Allergic reaction to procedure meds (General disorders) | 1
Amputation of treated limb above metatarsal line (General disorders) | 1
Amputation of treated limb below metatarsal line (General disorders) | 2
Artery perforation (General disorders) | 2
Death (General disorders) | 5
Dissection (General disorders) | 4
GI bleeding (General disorders) | 1
Hypotension (General disorders) | 1
Other Respiratory Issues (General disorders) | 1
Other Vascular Disorders (General disorders) | 1
Percutaneous revascularization of target vessel (General disorders) | 2
Renal Failure (General disorders) | 1
Restenosis (General disorders) | 64
Stent misplacement (General disorders) | 1
Stent/Vessel thrombosis (General disorders) | 4
Stroke (General disorders) | 1
Other (General disorders) | 15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EverFlex™ Peripheral Self-Expanding Stent System (N=287)
Angina (General disorders) | 17
Other Bleeding/lymphatic system disorders (General disorders) | 16
Other Cardiac Disorders (Cardiac disorders) | 24
Other Gastrointestinal Disorders (Gastrointestinal disorders) | 36
Other Infections (Infections and infestations) | 15
Other Musculoskeletal disorders (Musculoskeletal and connective tissue disorders) | 56
Other Vascular Disorders (Vascular disorders) | 65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less